CLINICAL TRIAL: NCT05359484
Title: Uroflowmetry Parameter (Delta Q Value) as a Noninvasive Tool to Discriminate Detrusor Underactivity From Bladder Outlet Obstruction
Brief Title: Delta Q Value to Discriminate Detrusor Underactivity From Bladder Outlet Obstruction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, principle investigator, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: K22/2019
Record Dates: First submitted 2022-04-23; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Urinary Obstruction; Detrusor Underactivity
MeSH Terms: conditions — Urinary Bladder, Underactive

STUDY DESIGN:
Intervention Model Description: Usage of Uroflowmetry to distinguish between bladder outlet obstruction and detrusor hypo-contractility
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- detrusor underactivity (Experimental): according to urodynamic, patients with weak urine stream were evaluated into 2 groups, either detrusor underactivity or bladder outflow obstruction From uroflowmetry, 5 variables including maximal flow rate (Qmax), average flow rate (Qave), voiding volume (VV), post void residual urine (PVR), and value of Qmax minus Qave (DeltaQ) were obtained.
  Interventions: Diagnostic Test: Uroflowmetry
- bladder out flow obstruction (Experimental): according to urodynamic, patients with weak urine stream were evaluated into 2 groups, either detrusor underactivity or bladder outflow obstruction From uroflowmetry, 5 variables including maximal flow rate (Qmax), average flow rate (Qave), voiding volume (VV), post void residual urine (PVR), and value of Qmax minus Qave (DeltaQ) were obtained.
  Interventions: Diagnostic Test: Uroflowmetry

INTERVENTIONS:
Diagnostic Test: Uroflowmetry — according to urodynamic, patients with weak urine stream were evaluated into 2 groups, either detrusor underactivity or bladder outflow obstruction From uroflowmetry, 5 variables including maximal flow rate (Qmax), average flow rate (Qave), voiding volume (VV), post-void residual urine (PVR), and value of Qmax minus Qaverage (DeltaQ) were obtained.

SUMMARY:
To determine the significance of delta Q value (Qmax - Qave) in discrimination between BOO and DU, to avoid invasive studies (pressure flow studies (PFSs)) and replace them with noninvasive study (uroflowmetry).

DETAILED DESCRIPTION:
lower urinary tract symptoms (LUTS) in old male patients are usually secondary to prostatic hyperplasia. However, it is becoming clear nowadays that prostatic enlargement is not always the cause of male LUTS, and other factors could cause male LUTS in the presence of benign prostate enlargement (BPE).

Two clinical situations are common in elderly patients like Bladder Outlet Obstruction (BOO) and Detrusor underactivity (DU) they affect the voiding phase in elderly men markedly.

To distinguish one from another may be challenging and could be only done by urodynamic study (UDS), which is the gold standard for diagnosis.

A urodynamic study is an invasive procedure, with side effects of pain and urinary tract infection, and the need for special equipment and expertise has limited its widespread use and made it very stressful for the patients.

On the other hand, Uroflowmetry is a non-invasive procedure that could be used in patients' assessments. A term of Delta Q is being used that focuses on the difference between (Qmax) and (Q-average). The hypothesis is that Delta Q would be lower in Detrusor underactivity because of the undermined detrusor function decreasing both average and maximum urine flow rate, but it is higher in BOO, which has normal detrusor contraction during the voiding phase.

Based on the concept uroflow can be used to replace urodynamic studies to differentiate between these 2 entities and hence to determine the proper management plan and to be a prognostic factor before surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* male patients aged over 50 years complaining of voiding symptoms
* International Prostatic Symptom Score (IPSS) 8 points or more,
* serum prostate-specific antigen (PSA) below 4 ng/ml
* no hematuria or pyuria.

Exclusion Criteria:

* Patients who were unable to complete the voiding study were deemed not eligible to participate in this review.
* patients with neurological causes of voiding dysfunction
* history of urinary tract abnormalities/lithiasis, lower urinary tract surgeries, urinary tract malignancy.
* acute UTI were excluded.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the main part of the bladder outlet obstruction is caused by the prostate that is why this study is based in male population
Enrollment: 238 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Q average | preoperative test, it is done only once and comparative evaluation with other parameters will be done
  Q average it represents the difference between Qmax and Q average in ml/sec as shown in uroflowmetry

SECONDARY OUTCOMES:
Q max | preoperative test, it is done only once and comparative evaluation with other parameters will be done
  uroflowmetry finding of maximum flow of urine in ml/sec
Q Average | preoperative test, it is done only once and comparative evaluation with other parameters will be done
  uroflowmetry finding of average flow of urine in ml/sec
post voiding residual urine | preoperative test, it is done only once and comparative evaluation with other parameters will be done
  amount of urine remains in the bladder after voiding as shown by Ultrasound in ml

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher, Cairo, Cairo Governorate, Egypt